CLINICAL TRIAL: NCT06821399
Title: Optimization and Evaluation of the Diagnosis and Treatment System for Diabetic Retinopathy in Type 2 Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: Yufan Wang (Other)
Responsible Party: Sponsor-Investigator, Yufan Wang, Chief Physician, Shanghai General Hospital, China
Organization: Shanghai General Hospital, China (Other)
Other Study IDs: 2023ZD0508104
Record Dates: First submitted 2025-01-02; First posted 2025-02-12 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Diabetes; Diabetic Retinopathy; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- DR High-Risk Population Cohort: An annual follow - up fundus examination is conducted. Metabolic differences are analyzed between the population with progressed diabetic retinopathy (DR) and those without progression. A predictive model for early warning of DR in type 2 diabetes is constructed to forecast the onset of DR one year later.
  Interventions: Diagnostic Test: Fundus Examination; Diagnostic Test: Metabolomics analysis
- Diabetic Retinopathy Early-Stage Population Cohort: Seeking specific metabolites that can reflect diabetic retinopathy and its severity in early - onset and late - onset type 2 diabetes mellitus (T2DM).
  Interventions: Diagnostic Test: Fundus Examination; Diagnostic Test: Metabolomics analysis
- Moderate-Stage Diabetic Retinopathy (DR) Population Cohort: Exploring a multidisciplinary model of chronic disease management for patients in the middle stage of diabetic retinopathy (DR), with both the endocrinology department and the ophthalmology department jointly developing standardized standard operating procedures for systemic and ocular examinations of metabolic diseases.
  Interventions: Diagnostic Test: Fundus Examination; Diagnostic Test: Metabolomics analysis
- Advanced-Stage Diabetic Retinopathy (DR) Population Cohort: The establishment of an integrated ward for diabetic eye diseases. For patients with severe diabetic eye diseases who urgently need ophthalmic surgery in the short term but have poor blood glucose control, the ophthalmology and endocrinology departments jointly manage and treat the patients. Endocrinologists adjust the blood glucose - lowering treatment plan. After the blood glucose stabilizes, ophthalmic surgery is performed. Continuous glucose monitoring is used to closely observe blood glucose fluctuations during the hospital stay, including intraoperative blood glucose. After the surgery, both ophthalmologists and endocrinologists jointly follow up with the patients.
  Interventions: Diagnostic Test: Fundus Examination; Diagnostic Test: Metabolomics analysis

INTERVENTIONS:
Diagnostic Test: Fundus Examination — Performing fundus photography on patients to assess the progression of diabetic retinopathy (DR).
Diagnostic Test: Metabolomics analysis — Conduct metabolomics testing at enrollment.

SUMMARY:
This study aims to integrate clinical indicators and features of fundus images, combined with metabolomics, to construct an early warning model for diabetic retinopathy (DR) in type 2 diabetes. By combining clinical indicators with metabolomics, the investigators aim to establish a precise DR typing model based on the age of diabetes onset (early-onset diabetes, late-onset diabetes) and based on the coexistence with two types of diabetic macrovascular complications. A multidisciplinary collaboration will be conducted for comprehensive management of DR to control the progression of moderate-stage DR. Cloud-based patient rooms combined with continuous glucose monitoring (CGM) will further explore the role of integrated diabetes retinopathy ward management models in the management of patients undergoing diabetes retinopathy surgery, pioneering a new model for the management of advanced DR.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for type 2 diabetes in the "China Type 2 Diabetes Prevention and Treatment Guidelines (2020 Edition)";

  * Aged between 20 and 79 years old, without other severe underlying diseases; ③ Possesses full cognitive and literacy abilities; ④ Volunteers to participate in this study and are willing to sign an informed consent form.

Exclusion Criteria:

* Those who have been diagnosed with type 1 or other types of diabetes;

  * Those with severe cardiac, pulmonary, hepatic, or renal insufficiency;

    * Those with mental confusion, speech disorders, or dementia, etc.;

      * Those who are unable to take care of themselves, bedridden, or have mobility impairments; ⑤ Women who are breastfeeding or pregnant;

        * Those with a recent history of surgery, trauma, acute major vascular complications, or infectious diseases.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetes Mellitus Patients
Sampling Method: Probability Sample
Enrollment: 2920 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Fundus examination | Conduct examinations at enrollment and twelve months after enrollment.
  Assess the severity of diabetic retinopathy (DR), and group accordingly. The high - risk DR cohort and the early - stage DR cohort have a fundus examination once a year; the mid - stage DR cohort has a fundus examination every six months; the late - stage DR cohort has a fundus examination every three months.

SECONDARY OUTCOMES:
Metabolomics analysis | at enrollment
  By metabolomics, we aim to establish a precise DR typing model based on the age of diabetes onset (early-onset diabetes, late-onset diabetes) and based on the coexistence with two types of diabetic macrovascular complications so that we can better prevent and treat diabetic retinopathy.
Triglycerides | Conduct examinations at enrollment, six months after enrollment, and twelve months after enrollment.
Glycated Hemoglobin | Conduct examinations at enrollment, six months after enrollment, and twelve months after enrollment.
Insulin levels | Conduct examinations at enrollment, six months after enrollment, and twelve months after enrollment.
Total Cholesterol | Conduct examinations at enrollment, six months after enrollment, and twelve months after enrollment.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The first hosptial of lanzhou university, Lanzhou
  - Shanghai general hosptial, Shanghai
  - The forth people's hosptial of shenyang, Shenyang